CLINICAL TRIAL: NCT05508009
Title: Phase 1b/2a Trial of Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) From an HLA-partially Matched Related or Unrelated Donor After TCRαβ+ T-cell/CD19+ B-cell Depletion for Patients Who Will Receive a Kidney Transplant (KT) From the Same HSCT/KT Donor
Brief Title: Early Trial of Allogeneic Hematopoietic Stem Cell Transplantation for Patients Who Will Receive a Kidney Transplant From the Same Donor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alice Bertaina (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor-Investigator, Alice Bertaina, Associate Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-65421
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: SIOD; Cystinosis; FSGS; SLE Nephritis; CKD Stage 4
MeSH Terms: conditions — Cystinosis; Lupus Nephritis | interventions — Cyclophosphamide; fludarabine; Whole-Body Irradiation; Rituximab; Melphalan; Kidney Transplantation

STUDY DESIGN:
Intervention Model Description: The study has two cohorts (Cohort 1b which will be safety lead-in with 4 patients, and then cohort 2a of 8 patients). The data generated will be compared with historical data available on outcomes of KT performed as SoC in this patient population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Cohort 1b: Conditioning Regimen A (Experimental): An initial cohort of 4 patients will be enrolled as part of the initial Phase 1b safety run-in evaluation. Patients will undergo an αβdepleted hematopoietic stem cell transplant (HSCT) after receiving conditioning regimen A (conditioning regimen type is dependent on underlying disease and not part of the experimental goals). In the presence of donor myeloid engraftment, at least 3 months post-HSCT, patients will undergo a living donor kidney transplant (KT) using same donor as HSCT. In the absence of any clinical signs of kidney rejection, pharmacological immunosuppression (used for KT) will be tapered off by Day +90 post-KT.
  Interventions: Drug: Cyclophosphamide 1200 mg/Kg; Drug: Fludarabine; Radiation: Total Body Irradiation; Drug: ATG; Drug: Rituximab; Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System; Procedure: Kidney Transplant
- Cohort 2a: Conditioning Regimen A (Experimental): If the intervention is determined to be safe and non-futile, the study will continue to enroll eight more patients under Phase 2a following the same treatment as Phase 1b.
  Interventions: Drug: Cyclophosphamide 1200 mg/Kg; Drug: Fludarabine; Radiation: Total Body Irradiation; Drug: ATG; Drug: Rituximab; Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System; Procedure: Kidney Transplant
- Cohort 1b: Conditioning Regimen B (Experimental): An initial cohort of 4 patients will be enrolled as part of the initial Phase 1b safety run-in evaluation. Patients will undergo an αβdepleted hematopoietic stem cell transplant (HSCT) after receiving conditioning regimen B (conditioning regimen type is dependent on underlying disease and not part of the experimental goals). In the presence of donor myeloid engraftment, at least 3 months post-HSCT, patients will undergo a living donor kidney transplant (KT) using same donor as HSCT. In the absence of any clinical signs of kidney rejection, pharmacological immunosuppression (used for KT) will be tapered off by Day +90 post-KT.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide 100 mg/Kg; Radiation: Total Body Irradiation; Drug: ATG; Drug: Rituximab; Drug: Melphalan; Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System; Procedure: Kidney Transplant
- Cohort 2a: Conditioning Regimen B (Experimental): If the intervention is determined to be safe and non-futile, the study will continue to enroll eight more patients under Phase 2a following the same treatment as Phase 1b.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide 100 mg/Kg; Radiation: Total Body Irradiation; Drug: ATG; Drug: Rituximab; Drug: Melphalan; Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System; Procedure: Kidney Transplant

INTERVENTIONS:
Drug: Cyclophosphamide 1200 mg/Kg — Cyclophosphamide 1200 mg/Kg will be administered as part of the conditioning regimen A prior to HSCT
  Arms: Cohort 1b: Conditioning Regimen A; Cohort 2a: Conditioning Regimen A
Drug: Fludarabine — Fludarabine (starting dose 0.5 mg/Kg and then PK guided to reach an AUC of 18-20) will be administered as part of the conditioning regimen prior to HSCT
Drug: Cyclophosphamide 100 mg/Kg — Cyclophosphamide 100 mg/Kg will be administered as part of the conditioning regimen B prior to HSCT
  Arms: Cohort 1b: Conditioning Regimen B; Cohort 2a: Conditioning Regimen B
Radiation: Total Body Irradiation — Total Body Irradiation 200 cGy will be administered as part of the conditioning regimen prior to HSCT
  Other Names: TBI
Drug: ATG — ATG 7.5 mg/Kg will be administered as part of the conditioning regimen prior to HSCT
Drug: Rituximab — Rituximab 200 mg/m2 will be administered within 24 hours of the HSCT
Drug: Melphalan — Melphalan 100 mg/m2 will be administered as part of the conditioning regimen prior to HSCT
  Arms: Cohort 1b: Conditioning Regimen B; Cohort 2a: Conditioning Regimen B
Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System — CliniMACS® TCRαβ-Biotin and CD19 Systems will be used to create the mobilized peripheral blood stem cells (PBSC) from allogeneic donors depleted of TCRαβ+ T cells and CD19+ B cells to be infused into the patient for the HSCT. The target dose for the number of CD34+ HSC infused is > 10 x 10^6 cells/Kg recipient weight. The minimum dose is 2 x 10^6 cells/Kg. There is no upper limit to the dose of CD34+ HSC infused as long as no more than 1 x 10^5 TCRαβ+ T-cells/Kg are infused. The target dose of TCRαβ+ T cells/Kg is < 0.50 x 10^5.
Procedure: Kidney Transplant — In the presence of donor myeloid engraftment, at least 3 months post-HSCT, with > 95% donor CD3+ chimerism, in the absence of signs of active aGvHD or cGvHD (moderate or severe), at least 4 weeks off of immunosuppression for any previously occurring acute or chronic GvHD (except single agent treatment of mild cGvHD), and with a BMI >18.5, ambulatory and active in addition to the eligibility for the standard of care KT criteria, patients will undergo a living donor KT using same donor as HSCT

SUMMARY:
This is a single center, non-randomized, non-controlled open-label phase 1b/2a trial of performing sequential αβdepleted-HSCT and KT in patients requiring KT to prevent kidney rejection post-KT, in the absence of any post-KT immunosuppression, to abrogate the need for lifelong immunosuppression, the risk of chronic rejection and, ultimately, the need for repeated transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated need for kidney transplant due to:

  a. Underlying genetic/immunologic disease the following conditions i. SIOD ii. FSGS iii. Cystinosis iv. SLE v. Membranoproliferative glomerulonephritis vi. Renal vasculitis characterized by positivity of the presence of ANCA vii. Other genetic diseases leading to kidney disease requiring KT Or b. Patients who have rejected a previous KT regardless of the underlying disease
* Chronic kidney disease (CKD) stage 3 or greater
* Steroids < 0.5 mg/Kg/day
* The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DQB1 and HLA-DRB1
* Lansky/Karnofsky score > 50; the Karnofsky Scale will be used in subjects ≥ 16 years of age, and the Lansky Scale will be used for those < 16 years of age.
* Able to give informed consent or have an LAR available to provide consent
* Male and female subjects of childbearing potential must agree to use an effective means of birth control to avoid pregnancy throughout the transplant procedure, while on immunosuppression, and if the subject experiences any cGvHD

Exclusion Criteria:

* Pregnant or lactating females.
* Greater than Grade II aGvHD or severe, unmanaged extensive cGvHD due to a previous allograft at the time of inclusion
* Dysfunction of liver (ALT/AST > 10 times upper normal value, or direct bilirubin > 3 times upper normal value), unmanageable dysfunction of renal function while undergoing dialysis
* Severe cardiovascular disease at the time of evaluation unresponsive to nutritional and dialytic support (left ventricular ejection fraction < 40%), or clinical or echocardiographic evidence of severe diastolic dysfunction
* Current active infectious disease. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load.
* Serious concurrent uncontrolled medical disorders except for primary disease leading to chronic kidney disease
* Lack of patient/parent/guardian informed consent
* Any severe concurrent disease which, in the judgement of the investigator would place the patient at increased risk during participation in the study

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2032-10 (Estimated); Study Completion 2034-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who are able to discontinue immunosuppression post-KT | Day +90 post-KT
  Donor chimerism equal or greater to 95% after successful HSCT/KT therapy allows for withdrawal of immunosuppressive therapy in patient

SECONDARY OUTCOMES:
Number of patients with successful kidney function | +1 year post-KT
  Normal renal function as measured by the glomerular filtration rate (GFR) using the CKiD Under 25 (U25) formula that includes the serum creatinine and the Cystatin C, along with normal protein excretion.
Number of patients with myloid engraftment | Day +42 post-HSCT
  Cumulative incidence of donor myeloid engraftment by Day +42 post-HSCT. Myeloid engraftment is defined as ANC of > 0.5 x 109/L for three consecutive laboratory values obtained on different days. Date of myeloid engraftment is the first date of the three lab values taken.
Number of patients with persistent full donor chimerism | Day +180 and 1 year post-KT
  >95% donor chimerism for myeloid and lymphoid cells as assessed by peripheral blood (total, CD15+, CD3+, CD19+, CD56+, and CD34+) chimerism by Short Tandem Repeat (STR) or next-generation sequencing (NGS) analysis
Number of patients with acute GvHD | Day +90 and Day +180 post-HSCT
  Cumulative incidence of acute GvHD (graded as II-IV and III-IV using the Magic criteria)
Number of patients with chronic GvHD | +1 year post-HSCT
  Cumulative incidence of chronic GvHD by NIH consensus criteria
Number of patients with de novo acute GVHD | +1 year post-KT
  Cumulative incidence of de novo acute GvHD (graded as II-IV and III-IV using the Magic criteria)
Number of patients with de novo chronic GVHD | +1 year post-KT
  Cumulative incidence of de novo chronic GVHD as measured by NIH consensus criteria
Number of patients with functional tolerance to donor cells | 6- and 12-months post-KT
  Lack of recipient immune response to donor cells when tested with mixed lymphocyte culture
Number of cases of secondary malignancies | +5 year post-KT
  New incidence of secondary malignancies in patients after study participation

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bertaina, MD, Principal Investigator — Stanford University; Paul Grimm, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dharnidharka VR, Fiorina P, Harmon WE. Kidney transplantation in children. N Engl J Med. 2014 Aug 7;371(6):549-58. doi: 10.1056/NEJMra1314376. No abstract available. PMID 25099579
- [Background] Poggio ED, Augustine JJ, Arrigain S, Brennan DC, Schold JD. Long-term kidney transplant graft survival-Making progress when most needed. Am J Transplant. 2021 Aug;21(8):2824-2832. doi: 10.1111/ajt.16463. Epub 2021 Feb 8. PMID 33346917
- [Background] Kawai T, Cosimi AB, Spitzer TR, Tolkoff-Rubin N, Suthanthiran M, Saidman SL, Shaffer J, Preffer FI, Ding R, Sharma V, Fishman JA, Dey B, Ko DS, Hertl M, Goes NB, Wong W, Williams WW Jr, Colvin RB, Sykes M, Sachs DH. HLA-mismatched renal transplantation without maintenance immunosuppression. N Engl J Med. 2008 Jan 24;358(4):353-61. doi: 10.1056/NEJMoa071074. PMID 18216355
- [Background] Kawai T, Sachs DH, Sprangers B, Spitzer TR, Saidman SL, Zorn E, Tolkoff-Rubin N, Preffer F, Crisalli K, Gao B, Wong W, Morris H, LoCascio SA, Sayre P, Shonts B, Williams WW Jr, Smith RN, Colvin RB, Sykes M, Cosimi AB. Long-term results in recipients of combined HLA-mismatched kidney and bone marrow transplantation without maintenance immunosuppression. Am J Transplant. 2014 Jul;14(7):1599-611. doi: 10.1111/ajt.12731. Epub 2014 Jun 5. PMID 24903438
- [Background] Kelter R. Bayesian Hodges-Lehmann tests for statistical equivalence in the two-sample setting: Power analysis, type I error rates and equivalence boundary selection in biomedical research. BMC Med Res Methodol. 2021 Aug 17;21(1):171. doi: 10.1186/s12874-021-01341-7. PMID 34404344
- [Background] Coemans M, Susal C, Dohler B, Anglicheau D, Giral M, Bestard O, Legendre C, Emonds MP, Kuypers D, Molenberghs G, Verbeke G, Naesens M. Analyses of the short- and long-term graft survival after kidney transplantation in Europe between 1986 and 2015. Kidney Int. 2018 Nov;94(5):964-973. doi: 10.1016/j.kint.2018.05.018. Epub 2018 Jul 24. PMID 30049474
- [Background] Lepeytre F, Dahhou M, Zhang X, Boucquemont J, Sapir-Pichhadze R, Cardinal H, Foster BJ. Association of Sex with Risk of Kidney Graft Failure Differs by Age. J Am Soc Nephrol. 2017 Oct;28(10):3014-3023. doi: 10.1681/ASN.2016121380. Epub 2017 Jun 7. PMID 28592422
- [Background] Kitchlu A, Dixon S, Dirk JS, Chanchlani R, Vasilevska-Ristovska J, Borges K, Dipchand AI, Ng VL, Hebert D, Solomon M, Michael Paterson J, Gupta S, Joseph Kim S, Nathan PC, Parekh RS. Elevated Risk of Cancer After Solid Organ Transplant in Childhood: A Population-based Cohort Study. Transplantation. 2019 Mar;103(3):588-596. doi: 10.1097/TP.0000000000002378. PMID 30048393
- [Background] Busque S, Scandling JD, Lowsky R, Shizuru J, Jensen K, Waters J, Wu HH, Sheehan K, Shori A, Choi O, Pham T, Fernandez Vina MA, Hoppe R, Tamaresis J, Lavori P, Engleman EG, Meyer E, Strober S. Mixed chimerism and acceptance of kidney transplants after immunosuppressive drug withdrawal. Sci Transl Med. 2020 Jan 29;12(528):eaax8863. doi: 10.1126/scitranslmed.aax8863. PMID 31996467
- [Background] Crompton KE, Elwood N, Kirkland M, Clark P, Novak I, Reddihough D. Feasibility of trialling cord blood stem cell treatments for cerebral palsy in Australia. J Paediatr Child Health. 2014 Jul;50(7):540-4. doi: 10.1111/jpc.12618. Epub 2014 Jun 9. PMID 24909743
- [Background] Scandling JD, Busque S, Lowsky R, Shizuru J, Shori A, Engleman E, Jensen K, Strober S. Macrochimerism and clinical transplant tolerance. Hum Immunol. 2018 May;79(5):266-271. doi: 10.1016/j.humimm.2018.01.002. Epub 2018 Jan 9. PMID 29330112
- [Background] Bertaina A, Merli P, Rutella S, Pagliara D, Bernardo ME, Masetti R, Pende D, Falco M, Handgretinger R, Moretta F, Lucarelli B, Brescia LP, Li Pira G, Testi M, Cancrini C, Kabbara N, Carsetti R, Finocchi A, Moretta A, Moretta L, Locatelli F. HLA-haploidentical stem cell transplantation after removal of alphabeta+ T and B cells in children with nonmalignant disorders. Blood. 2014 Jul 31;124(5):822-6. doi: 10.1182/blood-2014-03-563817. Epub 2014 May 28. PMID 24869942
- [Background] Bertaina A, Grimm PC, Weinberg K, Parkman R, Kristovich KM, Barbarito G, Lippner E, Dhamdhere G, Ramachandran V, Spatz JM, Fathallah-Shaykh S, Atkinson TP, Al-Uzri A, Aubert G, van der Elst K, Green SG, Agarwal R, Slepicka PF, Shah AJ, Roncarolo MG, Gallo A, Concepcion W, Lewis DB. Sequential Stem Cell-Kidney Transplantation in Schimke Immuno-osseous Dysplasia. N Engl J Med. 2022 Jun 16;386(24):2295-2302. doi: 10.1056/NEJMoa2117028. PMID 35704481